CLINICAL TRIAL: NCT04826627
Title: Association Between Preoperative Fasting, Intraoperative Glycemic Control, and Hospital Lenght of Stay in Children Younger Than 24 Months of Age Undergoing Scheduled Conventional Inpatient Surgery
Brief Title: Impact of Preoperative Fasting on Intraoperative Glycemic Homeostasis and Enhanced Recovery in Children
Acronym: GLYNEMCaen
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 19-041
Record Dates: First submitted 2021-03-31; First posted 2021-04-01 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2022-05

CONDITIONS: Anesthesia Morbidity; Child, Only; Fasting Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — Blood Glucose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: glycemia — capillary glycemia

SUMMARY:
In 2018, the main societies of anesthesia (European Society Anaesthesiology, European Society Pediatric Anesthesia, and Association des Anesthésistes Réanimateurs Pédiatriques d'Expression Française) changed the current recommendations for preoperative fasting time in children, reducing the time to last intake of clear liquids from two to one hour before anesthetic induction. Prolonged fasting may have a deleterious impact on blood glucose homeostasis. The consequences of intraoperative hypoglycemia in children can be serious in the short term, but also in the long term. The objective of multicenter prospective, observational cohort study is to investigate- in children younger than 24 months of age undergoing scheduled conventional inpatient surgery- a correlation between the duration of preoperative fasting, glycemic intraoperative homeostasis and the criteria of enhanced recovery after surgery, which are the hospital length of stay (main outcome), postoperative pain and postoperative nausea-vomiting (secondary outcomes). By identifying non-adherence to fasting rules as one of the causes of prolonged hospitalization, this study will highlight the need to develop effective strategies to promote adherence to fasting rules in pediatric surgery and minimize the potential deleterious impact on intraoperative glycemic control.

DETAILED DESCRIPTION:
Preoperative fasting instructions (6 hours for solids and formula, 4 hours for breast milk, and 1 hour for clear liquids) will be explained to parents orally during the preoperative anesthesia consultation and a written document, reminding them of these instructions, will be given to them afterwards.

Upon arrival in the operating room, the anesthesiologist will record on a standardized collection sheet the time of fasting as well as the premedication received (time of paracetamol and/or ibuprofen, β2-mimetic aerosols, preoperative antibiotic therapy).

After anesthetic induction, once airway management and securing of the peripheral venous line have been completed and before surgical setup, a capillary blood sample will be taken from the earlobe or fingertip to measure blood glucose and ketone levels using a blood glucose and ketone meter (FREESTYLE OPTIUM NEO H, ketone and blood sugar meter, calibration performed prior to the study by the pharmacology department). A ketonemia will be considered abnormally high if the ketone level is higher than 0.6 mmol/L (0.11g/L). Hypoglycemia will be defined as a capillary blood glucose level less than <3.5 mmol/L (0.63 g/L)9. In case of hypoglycemia or high ketonemia, a second capillary sample should be taken, taking care to change the sampling area (ear or finger) and then an average of the two results should be taken. Capillary blood glucose and ketone measurements are part of routine care in pediatric anesthesia. Therefore, there will be no additional cost.

Intraoperative monitoring for all children will include a 3-lead ECG, pneumocardiograph, non-invasive blood pressure measurement, pulse oximetry (SpO2), esophageal or rectal temperature measurement, and capnography. A forced-air heating blanket will be used to warm the patient during the procedure. Mean arterial pressure (MAP) will be documented after induction of anesthesia, and hypotension will be defined as MAP < 45 mmHg7. Intraoperatively, data will be collected from the patient's blood pressure.

Intraoperatively, the following data will be recorded on the standardized collection sheet: anesthetic agents used (hypnotics and morphinics), intraoperative analgesics, anti-nausea agents (dexamethasone, ondansetron), infusion fluids used (nature of the fluid, rate of infusion), catecholamine (ephedrine), drugs that may interfere with blood sugar regulation.

In the recovery room, postoperative pain will be evaluated using the EVENDOL scale and by the consumption of analgesics (total dose of paracetamol, ibuprofen, nalbuphine). The treatment of postoperative nausea and vomiting, left to the discretion of the anaesthetist, will also be recorded (total dose of ondansetron, droperidol, others).

After return to the department, the duration of hospitalization will be recorded. It will be defined as the number of days between arrival in the operating room and departure from the hospital. A clinically significant difference in length of stay will be considered a difference of at least 4 hours of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* All children less than 24 months of age
* scheduled for conventional inpatient surgery will be included

Exclusion Criteria:

* Children receiving intravenous fluids during the fasting period
* children managed in ambulatory surgery
* children with an ASA score strictly greater than 3
* children managed in the emergency operating room
* children with an acute metabolic disorder
* an endocrine pathology or a pathology requiring the chronic use of drugs modifying glycemia (insulin, oral antidiabetics, glucagon, gabapentin, antidepressants and neuroleptics, conversion enzyme inhibitors (CEI)
* beta blockers, statins, anti-transplant treatments, corticoids, antimalarial drugs, the following antibiotics fluoroquinolones, doxycycline, sulfamethoxazole, trimethoprim)

Ages: 0 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * All children less than 24 months of age
  * scheduled for conventional inpatient surgery will be included
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-04-14 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
length of stay in hospital | 1 week
  length of stay in hospital after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Caen Normandie, Caen
  - Hôpital Necker Enfants Malades, Paris